CLINICAL TRIAL: NCT05034653
Title: Cardiometabolic and Anthropometric Outcomes of Intermittent Fasting Among Overweight and Obese Civil Servants in Malaysia.
Brief Title: Intermittent Fasting Among Overweight and Obese Civil Servants in Malaysia.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ministry of Health, Malaysia (Other Government)
Responsible Party: Principal Investigator, Shazana Rifham binti Abdullah, Principle Investigator, Ministry of Health, Malaysia
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NMRR-19-3261-51726
Record Dates: First submitted 2021-08-23; First posted 2021-09-05 (Actual); Last update posted 2021-09-10 (Actual); Status verified 2021-09

CONDITIONS: Intermittent Fasting; Obesity
Keywords: Intermittent Fasting; Obesity; Overweight; Healthy Plate
MeSH Terms: conditions — Intermittent Fasting; Obesity; Overweight

STUDY DESIGN:
Intervention Model Description: This study applying mixed study method that consists of two parts: quantitative and qualitative. The quantitative part involved allocating participants into two intervention arms; combined Intermittent Fasting and Healthy Plate (IFHP) group and Healthy Plate (HP) group, and measuring the outcomes at baseline, 3-month and 6-month. On the other hand, the qualitative part aimed to explore the facilitators and barriers that enable or admonish the success of weight loss in the IFHP group through Focused Group Discussion that was conducted at month 6.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intermittent Fasting Healthy Plate (IFHP) (Experimental): Dry fasting from dawn to dusk for two days a week (Monday and Thursday) and Healthy Plate for the rest of the week. Female participants were discouraged from fasting during their menstruation period.
  Interventions: Other: Intermittent Fasting; Other: Healthy Plate
- Healthy Plate (Active Comparator): Practice the Healthy Plate concept in at least one meal every day
  Interventions: Other: Healthy Plate

INTERVENTIONS:
Other: Intermittent Fasting — During fasting day, no food or drink allowed from dawn to dusk
  Other Names: Dry Intermittent Fasting
  Arms: Intermittent Fasting Healthy Plate (IFHP)
Other: Healthy Plate — Quarter-quarter-half meal concept
  Other Names: Malaysian Healthy Plate

SUMMARY:
This study was a quasi-experimental study established to determine the cardio-metabolic, anthropometric, dietary intake and quality of life changes following combined Intermittent Fasting Healthy Plate and Healthy Plate interventions among overweight and obese civil servants.

DETAILED DESCRIPTION:
BACKGROUND

Overweight and obesity among adults is a growing global public health threat and an essential risk factor for various non-communicable diseases. Although it is largely preventable, the worldwide prevalence of obesity nearly tripled from 1975 and 2016 and remained increasing each year. In 2016, more than 1.9 billion adults were overweight, and 650 million were obese. If this current trend continues, it is estimated that 2.7 billion and over 1 billion adults will be overweight and obese by 2025, respectively.

Since obesity occurs due to positive energy balance in the body, the strategies of preventing and treating obesity mainly focus on dietary modification and increasing physical activity. One form of calorie restriction dietary protocol is intermittent fasting (IF), which encompasses various eating diet plans that cycle between a period of fasting and non-fasting over a defined period to create a negative energy balance, hence inducing weight loss. Studies have shown that IF is effective in reducing body weight and improving metabolic outcome. Although the effects of wet IF have been well documented, the benefits of dry IF (except for Ramadan fasting) is not clearly indicated in previous studies. Dry IF is defined as complete fasting without food and fluid intake.

As portion size is a crucial determinant of energy intake, portion control by controlling the serving size is another practical method to reduce calorie intake and promote weight loss. This portion control method has been widely practised and studied worldwide, using different portion divisions depends on the culture and eating habits. Malaysia Healthy Plate, a portion control dietary plan, was created to translate the messages in Malaysia Dietary Guideline 2010 and the Malaysia Food Pyramid 2010. It is a visual tool that emphasises the quarter-quarter-half concept that provides a quick visual technique that helps ensure the intake of food is within the recommended guideline. Specifically, Malaysia Healthy Plate is a single-meal guide that divides the plate into a quarter plate of grains or grains products, a quarter plate of fish, poultry, meat or egg, and a half plate of fruits and vegetables.

While weight losses are reported in studies of conventional IF, the adaptive phenomenon of dry IF on Monday and Thursday on cardiometabolic and anthropometric outcomes is still unclear. Similarly, although the policy of Malaysia Healthy Plate has been widely practised and publicised since 2010, the effectiveness of this eating plan in improving cardiometabolic risks and promoting weight loss is still not well documented. Thus, this study aimed to determine the cardiometabolic, anthropometric, dietary intake and quality of life changes among overweight and obese civil servants following combined Intermittent Fasting and Healthy Plate (IFHP) and Healthy Plate (HP), and to explore the participants' experience throughout the study. The investigators want to investigate whether combining dry IF and HP diet protocol will improve those parameters compared to HP alone.

METHODS

This was a mixed-method quasi-experimental study that evaluates the effectiveness of IFHP and HP among overweight and obese adults. A total of 177 participants were recruited in this study, of which 91 was allocated in the IFHP group and 86 in the HP group. The intervention comprises two phases; supervised (12 weeks) and unsupervised (12 weeks). The data collection was conducted during baseline, after the supervised phase (at week 12), and after the unsupervised phase (at week 24). For each participant, serum and whole blood were collected for analysis. Data on socio-demographic, quality of life, physical activity and dietary intake were also obtained using questionnaires during data collection.

The sample size calculation was conducted using the Power and Sample Size Program. It was followed the rules required for the comparison of two groups (10). The sample size was estimated using the level of significance (α =0.05) and power of the study (1-β=0.80), minimum suggested difference (delta) of 5% weight loss that may be achieved under this intervention and the corresponding differences between groups (SD=10%). The minimum sample size required for the study is 64 participants. By considering 40% attrition, the required sample size for each arm is 90 participants. The total number of participants required for this study is 180.

Data Management

To ascertain that the data collection and record-keeping are conducted efficiently, the Data Collection Booklet was developed and assigned to each participant of this study. This booklet consists of five sections (Socio-demographic, Quality of Life, Physical Activity, Dietary Record and Anthropometry Measurements Sections) sorted into three parts representing each point of data collection; baseline, month three and month six. This booklet was used as a data collection tool to record responses and measurements of the participant during baseline and follow-ups.

Data recorded in the booklet was then entered into a database at the end of the study. The data cleaning procedure was conducted by crosschecking all the entered data in the database and booklet and exploring the data to detect any significant outliers that possibly resulted from measurement error or data entering.

Data Analysis

Analysis was conducted using the Statistical Package of Social Science (SPSS) software version 25 (IBM Corp, NY). Data for continuous variables were presented by mean ± standard deviation (SD) or median and interquartile range (IQR) (for non-normally distributed data). For categorical variables, frequencies were calculated and presented together with percentages. Variables were compared using the independent t-test or Mann-Whitney U test for continuous variables and the Chi-squared or Fisher's exact (n≤5 in any cell) test for categorical variables. All statistical tests were two-sided and used a significance level of p <0.05. In further analysis, the repeated measures ANOVA will be used to compare the within and between groups changes of the outcomes.

ELIGIBILITY:
Inclusion Criteria:

* aged 19-59 years
* BMI of ≥ 23 kg/m2 (overweight or obese)
* who is ready to participate in the intervention (was assessed through readiness to participate screening)
* who can provide informed consent.

Exclusion Criteria:

* has recent involvement in weight loss program/activity (intermittent fasting/diet changes/physical activity changes or any activities that are performed constantly to reduce weight)
* suffering from any eating disorder
* was diagnosed with diabetes and hypertension (on medication) or other metabolic health disturbances such as thyroid disease, chronic kidney disease, malignancy and polycystic ovarian syndrome (PCOS)
* taking any medication or supplements that can affect study outcome
* pregnant
* has lack of capacity/language skills to independently follow the protocol were excluded from this study.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 177 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-04-07 (Actual); Study Completion 2021-05-05 (Actual)

PRIMARY OUTCOMES:
Body weight changes | Change from Baseline Body Weight at week 12
  Body weight changes measured in kilogram
Body weight changes | Change from Baseline Body Weight at week 24
  Body weight changes measured in kilogram
Body mass index (BMI) changes | Change from Baseline BMI at week 12
  Body mass index changes measured in kg/m^2 (weight in kilograms, height in meters)
Body mass index (BMI) changes | Change from Baseline BMI at week 24
  Body mass index changes measured in kg/m^2 (weight in kilograms, height in meters)
Waist-Hip Ratio (WHR) changes | Change from Baseline WHR at week 12
  WHR changes measured in centimeters (waist and hip circumference in centimeters)
Waist-Hip Ratio (WHR) changes | Change from Baseline WHR at week 24
  WHR changes measured in centimeters (waist and hip circumference in centimeters)
Body Fat Percentage changes | Change from Baseline Body Fat Percentage at week 12
  Body Fat Percentage changes measured in percentage
Body Fat Percentage changes | Change from Baseline Body Fat Percentage at week 24
  Body Fat Percentage changes measured in percentage
Body Fat Mass changes | Change from Baseline Body Fat Mass at week 12
  Body Fat Mass changes measured in kilograms
Body Fat Mass changes | Change from Baseline Body Fat Mass at week 24
  Body Fat Mass changes measured in kilograms
Fat Free Mass changes | Change from Baseline Body Fat Mass at week 12
  Fat Free Mass changes measured in kilograms
Fat Free Mass changes | Change from Baseline Body Fat Mass at week 24
  Fat Free Mass changes measured in kilograms
Systolic Blood Pressure changes | Change from Baseline Systolic Blood Pressure at week 12
  Systolic Blood Pressure changes measured in mmHg
Systolic Blood Pressure changes | Change from Baseline Systolic Blood Pressure at week 24
  Systolic Blood Pressure changes measured in mmHg
Diastolic Blood Pressure changes | Change from Baseline Diastolic Blood Pressure at week 12
  Diastolic Blood Pressure changes measured in mmHg
Diastolic Blood Pressure changes | Change from Baseline Diastolic Blood Pressure at week 24
  Diastolic Blood Pressure changes measured in mmHg
Fasting Blood Glucose changes | Change from Baseline Fasting Blood Glucose at week 12
  Fasting Blood Glucose changes measured in mmol/L
Fasting Blood Glucose changes | Change from Baseline Fasting Blood Glucose at week 24
  Fasting Blood Glucose changes measured in mmol/L
2-hour Post Prandial Blood Glucose changes | Change from Baseline 2-hour Post Prandial at week 12
  2-hour Post Prandial changes measured in mmol/L
2-hour Post Prandial Blood Glucose changes | Change from Baseline 2-hour Post Prandial at week 24
  2-hour Post Prandial changes measured in mmol/L
HbA1c changes | Change from Baseline HbA1c at week 12
  HbA1c changes measured in percentage
HbA1c changes | Change from Baseline HbA1c at week 24
  HbA1c changes measured in percentage
Fasting Total Cholesterol changes | Change from Baseline Fasting Total Cholesterol at week 12
  Fasting Total Cholesterol changes measured in mmol/L
Fasting Total Cholesterol changes | Change from Baseline Fasting Total Cholesterol at week 24
  Fasting Total Cholesterol changes measured in mmol/L
Fasting Triglyceride changes | Change from Baseline Fasting Triglyceride at week 12
  Fasting Triglyceride changes measured in mmol/L
Fasting Triglyceride changes | Change from Baseline Fasting Triglyceride at week 24
  Fasting Triglyceride changes measured in mmol/L
Fasting High-density Lipoprotein-Cholesterol (HDL-C) changes | Change from Baseline Fasting HDL-C at week 12
  Fasting HDL-C measured in mmol/L
Fasting High-density Lipoprotein-Cholesterol (HDL-C) changes | Change from Baseline Fasting HDL-C at week 24
  Fasting HDL-C measured in mmol/L
Fasting Low-density Lipoprotein-Cholesterol (LDL-C) changes | Change from Baseline Fasting LDL-C at week 12
  Fasting LDL-C measured in mmol/L
Fasting Low-density Lipoprotein-Cholesterol (LDL-C) changes | Change from Baseline Fasting LDL-C at week 24
  Fasting LDL-C measured in mmol/L
Fasting Insulin changes | Change from Baseline Fasting Insulin at week 12
  Fasting Insulin measured in uU/ml
Fasting Insulin changes | Change from Baseline Fasting Insulin at week 24
  Fasting Insulin measured in uU/ml

SECONDARY OUTCOMES:
Quality of Life changes | At baseline, week 12 and week 24
  Quality of Life score measured by Obesity and Weight-Loss Quality of Life (OWLQOL ) questionnaire
Dietary Intake changes | At baseline, week 12 and week 24
  Dietary intake changes measured by Food Frequency Questionnaire (FFQ)

CONTACTS AND LOCATIONS:
Locations (3):
- Malaysia (3):
  - National Institute of Health, Shah Alam, Selangor
  - Institut Latihan Kementerian Kesihatan Malaysia, Kuala Lumpur
  - Institute for Medical Research, Kuala Lumpur

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Abdullah SR, Azizul NH, Wan Mohd Zin RM, Sulaiman NS, Mustafa Khalid N, Mohd Salim Mullahi Jahn RJ, Khalil MKN, Abu Seman N, Zainal Abidin NA, Ali A, Tan YZ, Omar A, Johari MZ, Abdul Aziz NS, Baharudin A, Seman Z, Ibrahim Wong N, Md Rasip ML, Yusof HM, Md Noh MF. Cardiometabolic and Anthropometric Outcomes of Intermittent Fasting Among Civil Servants With Overweight and Obesity: Study Protocol for a Nonrandomized Controlled Trial. JMIR Res Protoc. 2022 Aug 5;11(8):e33801. doi: 10.2196/33801. PMID 35930331